CLINICAL TRIAL: NCT06591871
Title: Effect of Self-management Educational Program on Women's Self-care and Quality of Life Post Mastectomy Lymphedema
Brief Title: Educational Program on Self-Management for Women with Post-Mastectomy Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Ali Abd El-Rahman, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Lymphedema Post mastectomy
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post Mastectomy Lymphedema
Keywords: Post mastectomy lymphedema; Quality of life; Self-care; Self-management educational program
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Quasi-experimental research design was used for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Forty women with post-mastectomy lymphedema participated in this study. (Experimental): Forty women with post-mastectomy lymphedema participated in this study. All were free from other disabling conditions impeding self-care practices, hadn't previously received any educational programs about post-mastectomy lymphedema. The educational program was implemented through (5) sessions; (2 theoretical & 3 practical). Theoretical part included the following: a brief overview of anatomy and physiology of the lymphatic system, definition, causes, signs and symptoms, risk factors, stages, diagnosis and complications of post mastectomy lymphedema, also instructions about general practices for preventing and managing infection, hand and arm care, a healthy nutrition and when you call your physician. While, the practical part included the use of compression bandages, garments and their care, upper extremity lymphedema exercises and Manual Lymphatic Drainage (MLD) massage.
  Each session lasted 45 to 60 minutes and was conducted individually or in small groups of 2-3 women.
  Interventions: Other: Self-management educational program for post mastectomy lymphedema women

INTERVENTIONS:
Other: Self-management educational program for post mastectomy lymphedema women — The researcher created this program in response to the identified needs of post mastectomy lymphedema women to provide them with essential knowledge and self-care practices concerning post-mastectomy lymphedema. It was designed as a straightforward Arabic booklet written in simple language and supplemented with colorful illustrations and images to accommodate women of varying educational levels. It was consisted of two sections:
  Theoretical section included the following (A brief overview of anatomy and physiology of the lymphatic system, definition, causes, signs and symptoms, risk factors , stages, diagnosis and complications of post mastectomy lymphedema, also instructions about general practices for preventing and managing infection, hand and arm care ,a healthy nutrition and when you call your physician ).
  Practical section included (use of compression bandages, garments and their care, upper extremity lymphedema exercises, Manual Lymphatic Drainage (MLD) massage).

SUMMARY:
Post mastectomy lymphedema is a chronic disease that negatively affect physical, social, psychological and emotional well-being, so Patient education regarding self-management is crucial to enhance women's self -care and quality of life.

DETAILED DESCRIPTION:
Improvement in screening and treatment modalities of breast cancer has translated into higher survival rates in these patients. Unfortunately, this gain in survival leading to high prevalence of serious consequences of cancer treatments. Among these, post mastectomy lymphedema. It was estimated that 10 million women had breast cancer- related lymphedema (BCRL) worldwide, with 3-5 million affected in the United States. Approximately one in five women undergoing breast cancer surgery at risk for developing lymphedema .

Post-mastectomy lymphedema is a chronic and progressive tissue swelling caused by the abnormal buildup of protein-rich fluids in the interstitial space due to disrupted lymphatic drainage. This swelling results in physical symptoms such as heaviness, pain, decreased flexibility or tightness, stiffness, fatigue and numbness in the affected extremity. Its long-term burden extends beyond these physical symptoms, to significantly impact social, psychological, emotional functioning .also pose financial burdens to patients, the healthcare system, and society which lead to poor quality of life .

Lymphedema self-management constitutes the standard lymphedema treatment that should be maintained throughout life. In this context, the nurse's role becomes magnified. Self-management is the ability of individual to manage one's own chronic condition, encompassing the management of symptoms

, physical and psychosocial impacts, treatment, and incorporating these management practices into daily activities to attain optimal quality of life.

Nurses contribute significantly in management of post mastectomy lymphedema through educating the patients about lymphedema self-care behaviors which are important to control lymphedema symptoms, decrease lymphedema stages and prevent further progression of the disease. Lymphedema self-care involves maintaining risk-reduction behaviors, exercising, weight control, good nutrition, healthy lifestyle behaviors, caring and proper fit of compression garments, self-lymph drainage, skin care, signs and symptoms, preventing and managing infections.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with post-mastectomy lymphedema,free from other disabling conditions impeding self-care practices, No prior participation in lymphedema-related educational programs, and provided an agreement for participation in the study

Exclusion Criteria:

* Women with mental problems
* Unable to communicate with health team

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female with post mastectomy lymphedema
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Effect of self-management educational program on self-care of post mastectomy lymphedema women | three months
  Effect of self-management educational program on self-care of post mastectomy lymphedema women by using (The Breast Cancer Related Lymphedema (BCRL) Self-Care Scale). It comprised 31 items organized into four subdimensions called: Protection, activity and disease process management, pressure management, sustainability. Responses to these items were scored using a four-point likert scale: 4 for always, 3 for often, 2 for occasionally, and 1 for none. The scale yielded a minimum possible score of 31 and a maximum of 124.Higher scores reflect better self-care practices.

SECONDARY OUTCOMES:
Effect of self-management educational program on quality of life of post mastectomy lymphedema women | three months
  Effect of self-management educational program on quality of life of post mastectomy lymphedema women by using (Lymphedema Quality of Life Questionnaire-Arm (LYMQOL-Arm)).It comprises four domains with 21 questions and the last one about overall QoL. The domains are symptoms, appearance, function, and mood. Responses are evaluated on a four-point Likert scale: 1 (not at all), 2 (a little), 3 (quite a bit), and 4 (a lot). with higher scores indicating a worse QoL. Unlike the other questions, in question 21 (Q21) the patients are requested to rate their general quality of life from 0(poor)-10 (excellent). Higher scores of (Q21) indicate a better overall quality of life.
Effect of self-management educational program on knowledge of post mastectomy lymphedema women | three months
  Effect of self-management educational program on knowledge of post mastectomy lymphedema women by using Pre/Post Knowledge Assessment Questionnaire. It comprised two sections; first, an assessment of women's knowledge about post-mastectomy lymphedema, through nine multiple-choice questions (MCQs) .Second, knowledge regarding post mastectomy lymphedema self-care (10MCQs). Responses from these women were scored as one for each correct answer and zero for incorrect answers or unknown; the total score was calculated by summing the scores for all items and then transformed into a percentage. A percentage score of 60% or higher was considered satisfactory knowledge, while below 60% was considered unsatisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Ahmed, Dr, Study Director — Faculty of Nursing
Locations (1):
- faculty of nursing - Assiut University Hospital, Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donahue PMC, MacKenzie A, Filipovic A, Koelmeyer L. Advances in the prevention and treatment of breast cancer-related lymphedema. Breast Cancer Res Treat. 2023 Jul;200(1):1-14. doi: 10.1007/s10549-023-06947-7. Epub 2023 Apr 27. PMID 37103598